CLINICAL TRIAL: NCT01456923
Title: Phase 1 Study Of The Efficacy Of Chemotherapy With DNA Damaging Agents Versus Surgery In Colorectal Cancer
Brief Title: Chemotherapy With DNA Damaging Agents In Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centro Hospitalar Nordeste (Other)
Responsible Party: Principal Investigator, Ana Cadavez Pedro, Principal Investigator, Centro Hospitalar Nordeste
Purpose: Treatment
Other Study IDs: ACCRC10
Record Dates: First submitted 2011-10-18; First posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2008-09

CONDITIONS: Colorectal Cancer
Keywords: DNA damaging agents
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Therapeutics; Drug Therapy; Cohort Studies; Surgical Procedures, Operative

ARMS (2):
- Control (chemotherapy and surgery) (Active Comparator): Patients treated with chemotherapy + surgery
  Interventions: Other: Treatment with chemotherapy; Procedure: surgery
- Study (Active Comparator): Patients treated only with chemotherapy
  Interventions: Other: Only chemotherapy treatment for study cohort

INTERVENTIONS:
Other: Treatment with chemotherapy
  Arms: Control (chemotherapy and surgery)
Other: Only chemotherapy treatment for study cohort — Control patients were treated both with surgery and chemotherapy. Study patients were treated only with chemotherapy
  Arms: Study
Procedure: surgery
  Arms: Control (chemotherapy and surgery)

SUMMARY:
Chemotherapy Treatment alone with DNA damaging drugs might be as effective as chemotherapy combined with surgery in colorectal cancer (CRC) avoiding surgery complications.

ELIGIBILITY:
Inclusion Criteria:

- patients that did not underwent surgery

Exclusion Criteria:

- patients that underwent surgery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult